CLINICAL TRIAL: NCT05176483
Title: A Dose-Escalation and Expansion Study of the Safety and Efficacy of XL092 in Combination With Immuno-Oncology Agents in Subjects With Unresectable Advanced or Metastatic Solid Tumors
Brief Title: Study of Zanzalintinib in Combination With Immuno-Oncology Agents in Participants With Solid Tumors
Acronym: STELLAR-002
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL092-002; 2023-510061-10-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma (RCC); Metastatic Castration-Resistant Prostate Cancer (mCRPC); Urothelial Carcinoma (UC); Solid Tumor; Hepatocellular Carcinoma (HCC); Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Head and Neck Squamous Cell Carcinoma (HNSCC); Clear Cell Renal Cell Carcinoma (ccRCC); Non-Clear Cell Renal Cell Carcinoma (nccRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Ipilimumab; relatlimab

STUDY DESIGN:
Intervention Model Description: Dose-escalation followed by expansion phase with parallel assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Zanzalintinib + Nivolumab Dose-Escalation Cohorts (Experimental): Approximately 12 participants will accrue across 1-2 dose levels of Zanzalintinib following the "rolling 6" design.
  Interventions: Drug: Zanzalintinib; Drug: Nivolumab
- Zanzalintinib + Nivolumab + Ipilimumab Dose-Escalation Cohorts (Experimental): Approximately 12 participants will accrue across 1-2 dose levels of Zanzalintinib following the "rolling 6" design.
  Interventions: Drug: Zanzalintinib; Drug: Ipilimumab; Drug: Nivolumab
- Zanzalintinib + Nivolumab Expansion Cohorts (Experimental): The recommended dose from the dose-escalation stage may be further explored in tumor-specific cohorts.
  Interventions: Drug: Zanzalintinib; Drug: Nivolumab
- Zanzalintinib + Nivolumab + Ipilimumab Expansion Cohorts (Experimental): The recommended dose from the dose-escalation stage may be further explored in tumor-specific cohorts.
  Interventions: Drug: Zanzalintinib; Drug: Ipilimumab; Drug: Nivolumab
- Zanzalintinib Single-Agent Expansion Cohorts (Experimental)
  Interventions: Drug: Zanzalintinib
- Zanzalintinib + Nivolumab + Relatlimab Dose-Escalation Cohorts (Experimental): Approximately 12 participants will accrue across 1-2 dose levels of Zanzalintinib following the "rolling 6" design.
  Interventions: Drug: Zanzalintinib; Drug: Nivolumab + Relatlimab
- Zanzalintinib + Nivolumab + Relatlimab Expansion Cohorts (Experimental): The recommended dose from the dose-escalation stage may be further explored in tumor-specific cohorts.
  Interventions: Drug: Zanzalintinib; Drug: Nivolumab + Relatlimab

INTERVENTIONS:
Drug: Zanzalintinib — Zanzalintinib orally once daily (qd)
  Other Names: XL092
Drug: Nivolumab — 360 mg IV infusion once every 3 weeks (q3w)
  Other Names: Opdivo
  Arms: Zanzalintinib + Nivolumab Dose-Escalation Cohorts
Drug: Ipilimumab — 1 mg/kg IV infusion once every 3 weeks (q3w) for maximum of four doses
  Other Names: Yervoy
  Arms: Zanzalintinib + Nivolumab + Ipilimumab Dose-Escalation Cohorts; Zanzalintinib + Nivolumab + Ipilimumab Expansion Cohorts
Drug: Nivolumab — 3 mg/kg IV infusion once every 3 weeks (q3w) for first four doses, and then 480 mg IV infusion once every 4 weeks (q4w)
  Other Names: Opdivo
  Arms: Zanzalintinib + Nivolumab + Ipilimumab Dose-Escalation Cohorts; Zanzalintinib + Nivolumab + Ipilimumab Expansion Cohorts
Drug: Nivolumab — 480 mg IV infusion once every 4 weeks (q4w)
  Other Names: Opdivo
  Arms: Zanzalintinib + Nivolumab Expansion Cohorts
Drug: Nivolumab + Relatlimab — IV administration of nivolumab + relatlimab
  Arms: Zanzalintinib + Nivolumab + Relatlimab Dose-Escalation Cohorts; Zanzalintinib + Nivolumab + Relatlimab Expansion Cohorts

SUMMARY:
This is a multicenter Phase 1b, open label, dose-escalation and cohort-expansion study, evaluating the safety, tolerability, pharmacokinetics (PK), preliminary antitumor activity, and effect of biomarkers of zanzalintinib administered alone, and in combination with nivolumab (doublet), nivolumab + ipilimumab (triplet) and nivolumab + relatlimab (triplet) in participants with advanced solid tumors.

In the Expansion Stage, the safety and efficacy of zanzalintinib as monotherapy and in combination therapy will be further evaluated in tumor-specific Expansion Cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Cytologically or histologically confirmed solid tumor that is unresectable, locally advanced or metastatic.
* Dose-Escalation Cohorts: Participants with a solid tumor that is unresectable or metastatic and for which life-prolonging therapies do not exist or available therapies are intolerable or no longer effective.
* Expansion Cohort 1 (ccRCC): Participants with unresectable advanced or metastatic RCC with a clear cell component who have not received prior systemic therapy.

  * Note: Prior non-vascular endothelial growth factor (VEGF) targeted adjuvant or neoadjuvant is allowed if disease recurrence occurred 6 months after the last dose.
* Expansion Cohort 2 (ccRCC): Participants with unresectable advanced or metastatic RCC with a clear cell component.

  * Must have radiographically progressed after a combination therapy consisting of a Programmed Cell Death Protein 1 (PD-1)/Programmed death-ligand 1 (PD-L1) targeting monoclonal antibody (mAb) with a Vascular endothelial growth factor (receptor) tyrosine kinase inhibitor (VEGFR-TKI) or a PD-1 targeting mAb with a CTLA-4 mAb as the preceding line of therapy.
  * Must have received no more than one prior systemic anticancer therapy for unresectable advanced or metastatic renal cell carcinoma.
* Expansion Cohort 3 (mCRPC): Men with metastatic adenocarcinoma of the prostate.

  * Must have progressed during or after one novel hormone therapy (NHT) given for castration-sensitive locally advanced (T3 or T4) or metastatic castration-sensitive prostate cancer (CSPC), M0 CRPC, or mCRPC.
* Expansion Cohort 4 (UC, ICI-naive): Participants with histologically confirmed unresectable, locally advanced or metastatic transitional cell carcinoma of the urothelium (including the renal pelvis, ureter, urinary bladder, or urethra).

  * Must have progressed during or after prior first-line platinum-based combination therapy, including participants who received prior neoadjuvant or adjuvant platinum-containing therapy with disease recurrence < 12 months from the end of last therapy.
  * Must have received no more than 1 prior line of systemic anticancer therapy for unresectable, locally advanced or metastatic disease.
* Expansion Cohort 5 (post enfortumab vedotin [EV] and ICI): Participants with histologically confirmed unresectable, locally advanced or metastatic predominant urothelial carcinoma.

  * Progressive disease following prior EV or ineligible for EV, and progression following prior PD-1/PD-L1 inhibitor or ineligible for PD-1/PD-L1 inhibitor.
  * Prior receipt of platinum-based therapy allowed but not required.
  * Prior therapy with other agents allowed but not required.
* Expansion Cohort 6 (nccRCC): Participants with unresectable advanced or metastatic nccRCC of the following subtypes: Papillary, unclassified RCC, and translocation-associated, Fumarate Hydratase (FH) deficient and Succinate Dehydrogenase (SDH) deficient. Among the eligible histologic subtypes, sarcomatoid features are allowed.

  * No prior systemic anticancer therapy is allowed except adjuvant or neoadjuvant therapy if disease recurrence occurred at least 6 months after the last dose.
* Expansion Cohort 7 (HCC): Participants with locally advanced, or metastatic and/or unresectable HCC that is not amenable to curative treatment or locoregional therapy.
* Expansion Cohort 8 (NSCLC): Participants with Stage IV non-squamous NSCLC with positive PD-L1 expression (tumor proportion score [TPS] 1-49%) and without prior systemic anticancer therapy for metastatic disease.
* Expansion Cohort 9 (NSCLC): Participants with Stage IV non-squamous NSCLC who have radiologically progressed following treatment with one prior immune checkpoint inhibitor (anti-PD-1 or anti-PD-L1) for metastatic disease.
* Expansion Cohort 10 (CRC): Participants with histologically confirmed unresectable, locally advanced, or metastatic adenocarcinoma of the colon or rectum.
* Expansion Cohort 11 (HNSCC): Participant with inoperable, refractory, recurrent or metastatic HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx. PD-L1 combined positive score (CPS) ≥1.
* Expansion Cohort 12 (ccRCC): Participants with unresectable advance or metastatic RCC with a clear cell component, including participants who also have a sacromatoid feature.

  * Must have received no more than two prior lines of systemic anticancer therapy for unresectable advanced or metastatic renal cell carcinoma
* Expansion Cohort 13 and Cohort 14 (ccRCC 1L): Participants with unresectable advanced or metastatic RCC with a clear component, including participants who also have a sacromatoid feature.
* For all Expansion Cohorts except Cohort 3: Measurable disease per RECIST 1.1 as determined by the Investigator.
* For Expansion Cohorts 1 - 11 Only: Archival tumor tissue material, if available, or fresh tumor tissue if it can be safely obtained.
* Recovery to baseline or ≤ Grade 1 common terminology criteria for adverse events (CTCAE) v5 from AE(s) related to any prior treatments unless AE(s) are deemed clinically nonsignificant by the Investigator and/or stable on supportive therapy.
* Karnofsky Performance Status (KPS) ≥ 70%.
* Adequate organ and marrow function.
* Sexually active fertile participants and their partners must agree to use highly effective methods of contraception.
* Females of childbearing potential must not be pregnant at screening.

Key Exclusion Criteria:

* For all Dose-Escalation cohorts: Prior treatment with zanzalintinib. For all Expansion Cohorts: Prior treatment with zanzalintinib, nivolumab, ipilimumab or relatlimab with the following exceptions: Prior PD-1/PD-L1, Lymphocyte-activation gene 3 (LAG-3) and cCytotoxic T lymphocyte associated protein 4 (CTLA-4) targeting therapy for locally advanced or metastatic disease is allowed for Cohort 2 (ccRCC), Cohort 5 (UC), Cohort 9 (NSCLC), and Cohort 12 (ccRCC), and prior treatment in the neoadjuvant or adjuvant setting is allowed for Cohort 13 and Cohort 14 (ccRCC 1L).
* For all Dose-Escalation Cohorts and Expansion Cohort 2 (ccRCC), 3 (mCRPC), Cohort 5 (UC), Cohort 9 (NSCLC), Cohort 10 (CRC), and Cohort 12: Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* For Cohort 3 (mCRPC): Receipt of abiraterone within 1 week; cyproterone within 10 days; or receipt of flutamide, nilutamide, bicalutamide, enzalutamide, or other androgen receptor inhibitors within 2 weeks before first dose of study treatment.
* For all Dose-Escalation Cohorts and Expansion Cohort 2 (ccRCC), Cohort 3 (mCRPC), Cohort 5 (UC), Cohort 9 (NSCLC) and Cohort 10 (CRC), and Cohort 12: Receipt of any type of anticancer antibody or systemic chemotherapy within 4 weeks before first dose of study treatment.
* Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks before first dose of study treatment.
* Prior external radiation therapy for bone metastasis within 2 weeks, for other tumor sites within 4 weeks, and prior radium-223 therapy within 6 weeks before first dose of study treatment, unless otherwise specified.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.
* Concomitant anticoagulation with oral anticoagulants, except for specified direct factor Xa inhibitors.
* Administration of a live, attenuated vaccine within 30 days prior to first dose.
* Uncontrolled, significant intercurrent or recent illness.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 460 ms for females and > 450 ms for males per electrocardiogram (ECG) within 14 days before first dose of study treatment.
* Participants with inadequately treated adrenal insufficiency.
* Pregnant or lactating females.
* Any other active malignancy within two years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy. Incidentally diagnosed prostate cancer is allowed if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6.
* For Cohort 2 (ccRCC, 2L): Receipt of a prior triplet therapy including a VEGFR-TKI, a PD1 targeting mAb, and a CTLA-4 mAb.
* For Cohort 3 (mCRPC): Receipt of a taxane-based chemotherapy for mCRPC.
* For Cohort 4 (UC, ICI-naïve): Participants who have had recurrence within the 6 months of completing adjuvant anti-PD-(L)1 treatment.
* For Cohort 6 (nccRCC, 1L): Participants with chromophobe, renal medullary carcinoma, or pure collecting duct nccRCC.
* For Cohort 7 (HCC):

  * Documented hepatic encephalopathy (HE) within 6 months before the first dose.
  * Clinically meaningful ascites (ie, ascites requiring paracentesis or escalation in diuretics) within 6 months before randomization.
  * Participants who have received any local anticancer therapy including surgery, percutaneous ethanol injection (PEI), radiofrequency ablation (RFA), microwave ablation (MWA), transarterial chemoembolization (TACE), or transarterial radioembolization (TARE) within 28 days prior to first dose.
  * Participants with known fibrolamellar carcinoma, sarcomatoid HCC, or mixed hepatocellular cholangiocarcinoma
* For Cohort 10 (CRC, 2L+): Receipt of prior therapy with regorafenib and/or trifluridine + tipiracil (TAS-102).
* For Cohort 11 (HNSCC): Primary tumor site of the nasopharyngeal area.
* For Cohorts 1 (ccRCC, 1L), 2 (ccRCC, 2L), 4, 5 (UC), 7 (HCC), 8 (NSCLC 1L PD-L1 low), 9 (NSCLC, 2L+), 10 (CRC, microsatellite stable [MSS], 2L+), and 11 (HNSCC):

  * Troponin T (TnT) or I (TnI) > 2 × institutional upper limit of normal (ULN).

Note: Additional Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2030-06-28 (Estimated); Study Completion 2030-06-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs), Including Immune-Mediated Adverse Events (imAEs) | Up to 36 months
Expansion Stage: Objective Response Rate (ORR) | Up to 24 months
  To evaluate ORR in participants with measurable disease as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors guideline version 1.1 (RECIST 1.1).
Expansion Stage Cohort 3 (mCRPC): Progression-Free Survival (PFS) | Up to 24 months
  To evaluate duration of radiographic PFS as determined per Prostate Working Group 3 (PCWG3) criteria by Blinded Independent Radiology Committee (BIRC).
Expansion Stage Cohort 10 (CRC): Overall Survival (OS) | 6 months

SECONDARY OUTCOMES:
Expansion Stage: Duration of Response (DOR) | Up to 24 months
  To evaluate DOR in participants with measurable disease as assessed by the Investigator per RECIST 1.1.
Expansion Stage: Progression-Free Survival (PFS) | Up to 24 months
  To evaluate PFS in participants with measurable disease as assessed by the Investigator per RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (122):
- United States (46):
  - Exelixis Clinical Site #67, Phoenix, Arizona
  - Exelixis Clinical Site #1, Tucson, Arizona
  - Exelixis Clinical Site #123, Palo Alto, California
  - Exelixis Clinical Site #59, Santa Barbara, California
  - Exelixis Clinical Site #87, Littleton, Colorado
  - Exelixis Clinical Site #62, New Haven, Connecticut
  - Exelixis Clinical Site #49, Newark, Delaware
  - Exelixis Clinical Site #48, Celebration, Florida
  - Exelixis Clinical Site #11, Gainesville, Florida
  - Exelixis Clinical Site #78, Jacksonville, Florida
  - Exelixis Clinical Site #47, Miami, Florida
  - Exelixis Clinical Site #61, Plantation, Florida
  - Exelixis Clinical Site #8, Tampa, Florida
  - Exelixis Clinical Site #26, Chicago, Illinois
  - Exelixis Clinical Site #4, Indianapolis, Indiana
  - Exelixis Clinical Site #122, Louisville, Kentucky
  - Exelixis Clinical Site #14, Baltimore, Maryland
  - Exelixis Clinical Site #7, Boston, Massachusetts
  - Exelixis Clinical Site #65, Detroit, Michigan
  - Exelixis Clinical Site #13, Detroit, Michigan
  - Exelixis Clinical Site #68, Rochester, Minnesota
  - Exelixis Clinical Site #2, Omaha, Nebraska
  - Exelixis Clinical Site #5, Omaha, Nebraska
  - Exelixis Clinical Site #55, Las Vegas, Nevada
  - Exelixis Clinical Site #88, East Brunswick, New Jersey
  - Exelixis Clinical Site #105, Hackensack, New Jersey
  - Exelixis Clinical Site #60, New York, New York
  - Exelixis Clinical Site #6, New York, New York
  - Exelixis Clinical Site #76, Syracuse, New York
  - Exelixis Clinical Site #12, Durham, North Carolina
  - Exelixis Clinical Site #10, Cleveland, Ohio
  - Exelixis Clinical Site #51, Portland, Oregon
  - Exelixis Clinical Site #104, Hershey, Pennsylvania
  - Exelixis Clinical Site #98, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #32, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #24, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #9, Myrtle Beach, South Carolina
  - Exelixis Clinical Site #3, Nashville, Tennessee
  - Exelixis Clinical Site #46, Austin, Texas
  - Exelixis Clinical Site #111, Dallas, Texas
  - Exelixis Clinical Site #89, Dallas, Texas
  - Exelixis Clinical Site #73, Irving, Texas
  - Exelixis Clinical Site #50, Plano, Texas
  - Exelixis Clinical Site #70, Tyler, Texas
  - Exelixis Clinical Site #66, Charlottesville, Virginia
  - Exelixis Clinical Site #33, Milwaukee, Wisconsin
- Australia (5):
  - Exelixis Clinical Site #116, Albury
  - Exelixis Clinical Site #35, Birtinya
  - Exelixis Clinical Site #16, Brisbane
  - Exelixis Clinical Site #42, Saint Leonards
  - Exelixis Clinical Site #36, Sydney
- Austria (4):
  - Exelixis Clinical Site #94, Graz
  - Exelixis Clinical Site #31, Salzburg
  - Exelixis Clinical Site #29, Vienna
  - Exelixis Clinical Site #106, Wein
- Belgium (2):
  - Exelixis Clinical Site #39, Anderlecht
  - Exelixis Clinical Site #37, Kortrijk
- France (14):
  - Exelixis Clinical Site #85, Besançon
  - Exelixis Clinical Site #96, Bordeaux
  - Exelixis Clinical Site #79, Caen
  - Exelixis Clinical Site #118, Clermont-Ferrand
  - Exelixis Clinical Site #109, Lyon
  - Exelixis Clinical Site #92, Marseille
  - Exelixis Clinical Site #64, Nice
  - Exelixis Clinical Site #83, Paris
  - Exelixis Clinical Site #91, Paris
  - Exelixis Clinical Site #80, Rennes
  - Exelixis Clinical Site #63, Saint-Herblain
  - Exelixis Clinical Site #75, Strasbourg
  - Exelixis Clinical Site #84, Vandœuvre-lès-Nancy
  - Exelixis Clinical Site #115, Villejuif
- Germany (9):
  - Exelixis Clinical Site #103, Essen
  - Exelixis Clinical Site #113, Hamburg
  - Exelixis Clinical Site #108, Heidelberg
  - Exelixis Clinical Site #82, Herne
  - Exelixis Clinical Site #93, Jena
  - Exelixis Clinical Site #112, München
  - Exelixis Clinical Site #102, Nürtingen
  - Exelixis Clinical Site #107, Trier
  - Exelixis Clinical Site #95, Tübingen
- Israel (6):
  - Exelixis Clinical Site #86, Beersheba
  - Exelixis Clinical Site #72, Haifa
  - Exelixis Clinical Site #52, Jerusalem
  - Exelixis Clinical Site #71, Petah Tikva
  - Exelixis Clinical Site #69, Tel Aviv
  - Exelixis Clinical Site #38, Ẕerifin
- Italy (7):
  - Exelixis Clinical Site #121, Ancona
  - Exelixis Clinical Site #117, Bologna
  - Exelixis Clinical Site #90, Florence
  - Exelixis Clinical Site #101, Milan
  - Exelixis Clinical Site #81, Milan
  - Exelixis Clinical Site #40, Napoli
  - Exelixis Clinical Site #74, Ravenna
- New Zealand (2):
  - Exelixis Clinical Site #30, Grafton
  - Exelixis Clinical Site #45, Hamilton
- Poland (5):
  - Exelixis Clinical Site #20, Bydgoszcz
  - Exelixis Clinical Site #28, Gdansk
  - Exelixis Clinical Site #34, Otwock
  - Exelixis Clinical Site #54, Poznan
  - Exelixis Clinical Site #114, Wroclaw
- Spain (16):
  - Exelixis Clinical Site #41, Badajoz
  - Exelixis Clinical Site #53, Barcelona
  - Exelixis Clinical Site #15, Barcelona
  - Exelixis Clinical Site #27, Barcelona
  - Exelixis Clinical Site #120, L'Hospitalet de Llobregat
  - Exelixis Clinical Site #57, Madrid
  - Exelixis Clinical Site #43, Madrid
  - Exelixis Clinical Site #58, Madrid
  - Exelixis Clinical Site #77, Madrid
  - Exelixis Clinical Site #19, Madrid
  - Exelixis Clinical Site #100, Madrid
  - Exelixis Clinical Site #18, Pamplona
  - Exelixis Clinical Site #119, Santander
  - Exelixis Clinical Site #23, Seville
  - Exelixis Clinical Site #56, Valencia
  - Exelixis Clinical Site #25, Valencia
- Switzerland (3):
  - Exelixis Clinical Site #21, Chur
  - Exelixis Clinical Site #22, Sankt Gallen
  - Exelixis Clinical Site #44, Winterthur
- United Kingdom (3):
  - Exelixis Clinical Site #110, Cambridge
  - Exelixis Clinical Site #99, London
  - Exelixis Clinical Site #97, Middlesex

IPD SHARING:
Plan to Share IPD: No